CLINICAL TRIAL: NCT00014001
Title: Comparative Effectiveness of Antipsychotic Medications in Patients With Schizophrenia (CATIE Schizophrenia Trial)
Brief Title: CATIE- Schizophrenia Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH090001-06; N01MH90001-SZ; DSIR AT; N01MH90001 (NIH); N01MH090001 (NIH)
Record Dates: First submitted 2001-04-06; First posted 2001-04-09 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2006-10

CONDITIONS: Schizophrenia
Keywords: Antipsychotic Treatment; Effectiveness
MeSH Terms: conditions — Schizophrenia | interventions — Perphenazine; Olanzapine; Quetiapine Fumarate; Risperidone; ziprasidone; Clozapine; fluphenazine depot

INTERVENTIONS:
Drug: perphenazine
Drug: olanzapine
Drug: quetiapine
Drug: risperidone
Drug: ziprasidone
Drug: clozapine
Drug: fluphenazine decanoate

SUMMARY:
The CATIE Schizophrenia Trial is part of the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Project. The schizophrenia trial is being conducted to determine the long-term effects and usefulness of antipsychotic medications in persons with schizophrenia. It is designed for people with schizophrenia who may benefit from a medication change. The study involves the newer atypical antipsychotics (olanzapine, quetiapine, risperidone, clozapine, and ziprasidone)and the typical antipsychotics (perphenazine and fluphenazine decanoate). All participants will receive an initial comprehensive medical and psychiatric evaluation and will be closely followed throughout the study. For most participants the study will last up to 18 months. Everyone in the study will be offered an educational program about schizophrenia and family members will be encouraged to participate.

DETAILED DESCRIPTION:
This trial will consist of 1600 patients with schizophrenia for whom a medication change may be indicated for reasons of limited efficacy or tolerability. All patients will receive some psychosocial treatment through study participation. Research participants and their family members will be offered psychosocial interventions directed at improving patient and family understanding of the illness, decreasing the burden of illness in the family, maximizing treatment adherence, minimizing relapse, enhancing access to a range of community-based rehabilitative services and improving study retention.

Phase I: Patients will be randomly assigned to one of five treatment conditions for up to 18 months:

1. 320 begin double-blind treatment with perphenazine (PER)
2. 320 begin double-blind treatment with olanzapine (OLZ)
3. 320 begin double-blind treatment with quetiapine (QUET)
4. 320 begin double-blind treatment with risperidone (RIS)
5. 220 begin double-blind treatment with ziprasidone (ZIP)

Phase IA: 100 patients screened and found to have tardive dyskinesia who would otherwise be eligible for the study will be randomly assigned to one of the four atypical drugs in Phase IA.

Phase IB: Patients who fail treatment with perphenazine in Phase I will be randomly assigned to olanzapine, quetiapine, or risperidone in Phase IB.

Phase II: Patients who discontinue their initial assigned atypical antipsychotic treatment in Phase I, IA, or IB for any non-administrative reason will proceed to their second assigned treatment (third for Phase IB patients) and will be followed for up to the remainder of their 18-month participation, as follows:

1. Patients originally assigned to one of the newer atypical antipsychotics who discontinue due to efficacy failure will be randomly assigned to double-blind treatment with one of the other two newer atypical antipsychotics (OLZ, RIS, QUET) which they had not previously received (50%) or with open label clozapine (50%).
2. Patients originally assigned to one of the newer atypical antipsychotics who discontinue due to tolerability failure will be randomly assigned to double-blind treatment with one of the other newer atypical antipsychotics (OLZ, RIS, QUET) which they had not previously received (50%), or with ziprasidone (50%). Until ziprasidone is activated, all patients will be assigned to one of the other atypical antipsychotics.

Phase II will last at least 6 months, even if that means participants stay in the study for more than 18 months

Phase III: Patients who discontinue Phase II will be recommended open treatment with the preferred regimen based on their treatment history in the study. The treatment options include clozapine, newer atypical antipsychotic (olanzapine, risperidone, quetiapine, ziprazidone, and aripiprazole), fluphenazine decanoate, perphenazine, and dual antipsychotic therapy using two of these drugs.

Note: All treatments will be double-blinded in treatment Phases I and II except for clozapine.

ELIGIBILITY:
Inclusion

* 18-65 years old
* DSM-IV diagnosis of schizophrenia
* adequate capacity to consent

Exclusion

* Intolerance or failure to respond to one of the treatments
* Diagnoses of schizoaffective disorder, mental retardation, pervasive developmental disorder, delirium, dementia, amnesia
* First episode of schizophrenia
* Women currently pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2000-12; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Study Director — University of North Carolina
Locations (54):
- United States (54):
  - Synergy Clinical Research, Chula Vista, California
  - LA County-University of Southern California Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California,San Diego/VA Medical System, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Harbor UCLA Research & Education Institute, Torrance, California
  - New Britain General Hospital, New Britain, Connecticut
  - Yale University/Connecticut Mental Health Center, New Haven, Connecticut
  - Mental Health Advocates Inc., Boca Raton, Florida
  - VA Medical Center, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Medical School Department of Psychiatry, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Psychiatric Research Institute, Outpatient Clinic, Wichita, Kansas
  - Louisiana State University Health Services Center, Shreveport, Louisiana
  - Clinical Insights, Inc., Glen Burnie, Maryland
  - Massachusetts General Hospital-Freedom Trial Clinic Schizophrenia Program, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Corrigan Mental Health Center, Fall River, Massachusetts
  - University Of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Minnesota School of Medicine, Minneapolis, Minnesota
  - University of Mississippi VA Medical Center, Jackson, Mississippi
  - University of Missouri Kansas City Medical School, Kansas City, Missouri
  - Burrell Behavioral Health-Cox North Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albuquerque VA Medical Center, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Mount Sinai Medical Center-Bronx VA Medical Center, The Bronx, New York
  - Duke University Medical Center-John Umstead Hospital, Butner, North Carolina
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Behavioral Health Center, Charlotte, North Carolina
  - Dorothea Dix Hospital, Raleigh, North Carolina
  - Appalachian Psychiatric Healthcare System, Athens, Ohio
  - North East Ohio Health Services, Beachwood, Ohio
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Eastern Pennsylvania Psychiatric Institute, Philadelphia, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center, Charleston, South Carolina
  - Vanderbilt University Schizophrenia Research, Nashville, Tennessee
  - Tri-County MHMR Services, Conroe, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Life Management Center for MH/MR Services, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - MHMRA of Harris County-Northwest Community Service Center, Houston, Texas
  - The Center for Health Care Services, San Antonio, Texas
  - Valley Mental Health Psychopharmacology Research Center, Salt Lake City, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Tacoma, Washington

REFERENCES:
- [Background] Davis SM, Koch GG, Davis CE, LaVange LM. Statistical approaches to effectiveness measurement and outcome-driven re-randomizations in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) studies. Schizophr Bull. 2003;29(1):73-80. doi: 10.1093/oxfordjournals.schbul.a006993. PMID 12908662
- [Background] Keefe RS, Mohs RC, Bilder RM, Harvey PD, Green MF, Meltzer HY, Gold JM, Sano M. Neurocognitive assessment in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) project schizophrenia trial: development, methodology, and rationale. Schizophr Bull. 2003;29(1):45-55. doi: 10.1093/oxfordjournals.schbul.a006990. PMID 12908660
- [Background] Lieberman JA, Stroup TS. Guest editors' introduction: what can large pragmatic clinical trials do for public mental health care? Schizophr Bull. 2003;29(1):1-6. doi: 10.1093/oxfordjournals.schbul.a006979. No abstract available. PMID 12908656
- [Background] Rosenheck R, Doyle J, Leslie D, Fontana A. Changing environments and alternative perspectives in evaluating the cost-effectiveness of new antipsychotic drugs. Schizophr Bull. 2003;29(1):81-93. doi: 10.1093/oxfordjournals.schbul.a006994. PMID 12908663
- [Background] Sernyak MJ, Leslie D, Rosenheck R. Use of system-wide outcomes monitoring data to compare the effectiveness of atypical neuroleptic medications. Am J Psychiatry. 2003 Feb;160(2):310-5. doi: 10.1176/appi.ajp.160.2.310. PMID 12562578
- [Background] Stroup TS, McEvoy JP, Swartz MS, Byerly MJ, Glick ID, Canive JM, McGee MF, Simpson GM, Stevens MC, Lieberman JA. The National Institute of Mental Health Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) project: schizophrenia trial design and protocol development. Schizophr Bull. 2003;29(1):15-31. doi: 10.1093/oxfordjournals.schbul.a006986. PMID 12908658
- [Background] Swartz MS, Perkins DO, Stroup TS, McEvoy JP, Nieri JM, Haak DC. Assessing clinical and functional outcomes in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia trial. Schizophr Bull. 2003;29(1):33-43. doi: 10.1093/oxfordjournals.schbul.a006989. PMID 12908659
- [Background] Stroup TS, Appelbaum PS. Evaluation of "subject advocate" procedures in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia study. Schizophr Bull. 2006 Jan;32(1):147-52. doi: 10.1093/schbul/sbj026. Epub 2005 Nov 10. PMID 16282635
- [Result] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Result] McEvoy JP, Lieberman JA, Stroup TS, Davis SM, Meltzer HY, Rosenheck RA, Swartz MS, Perkins DO, Keefe RS, Davis CE, Severe J, Hsiao JK; CATIE Investigators. Effectiveness of clozapine versus olanzapine, quetiapine, and risperidone in patients with chronic schizophrenia who did not respond to prior atypical antipsychotic treatment. Am J Psychiatry. 2006 Apr;163(4):600-10. doi: 10.1176/ajp.2006.163.4.600. PMID 16585434
- [Result] Stroup TS, Lieberman JA, McEvoy JP, Swartz MS, Davis SM, Rosenheck RA, Perkins DO, Keefe RS, Davis CE, Severe J, Hsiao JK; CATIE Investigators. Effectiveness of olanzapine, quetiapine, risperidone, and ziprasidone in patients with chronic schizophrenia following discontinuation of a previous atypical antipsychotic. Am J Psychiatry. 2006 Apr;163(4):611-22. doi: 10.1176/ajp.2006.163.4.611. PMID 16585435
- [Result] Rosenheck RA, Leslie DL, Sindelar J, Miller EA, Lin H, Stroup TS, McEvoy J, Davis SM, Keefe RS, Swartz M, Perkins DO, Hsiao JK, Lieberman J; CATIE Study Investigators. Cost-effectiveness of second-generation antipsychotics and perphenazine in a randomized trial of treatment for chronic schizophrenia. Am J Psychiatry. 2006 Dec;163(12):2080-9. doi: 10.1176/ajp.2006.163.12.2080. PMID 17151158
- [Result] Essock SM, Covell NH, Davis SM, Stroup TS, Rosenheck RA, Lieberman JA. Effectiveness of switching antipsychotic medications. Am J Psychiatry. 2006 Dec;163(12):2090-5. doi: 10.1176/ajp.2006.163.12.2090. PMID 17151159
- [Derived] Fabbri C, Leggio GM, Drago F, Serretti A. Imputed expression of schizophrenia-associated genes and cognitive measures in patients with schizophrenia. Mol Genet Genomic Med. 2022 Jun;10(6):e1942. doi: 10.1002/mgg3.1942. Epub 2022 Apr 30. PMID 35488718
- [Derived] Beaudoin M, Hudon A, Giguere CE, Potvin S, Dumais A. Prediction of quality of life in schizophrenia using machine learning models on data from Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia trial. Schizophrenia (Heidelb). 2022 Mar 21;8(1):29. doi: 10.1038/s41537-022-00236-w. PMID 35314708
- [Derived] Miller BJ, McEvoy JP, McCall WV. Insomnia, Suicidal Ideation, and Suicide Attempts in the Clinical Antipsychotic Trials of Intervention Effectiveness. J Clin Psychiatry. 2021 Mar 23;82(3):20m13338. doi: 10.4088/JCP.20m13338. PMID 34033271
- [Derived] Pathak S, Jiang Y, DiPetrillo L, Todtenkopf MS, Liu Y, Correll CU. Course of Psychosis in Schizophrenia With Alcohol Use Disorder: A Post Hoc Analysis of the Clinical Antipsychotic Trials of Intervention Effectiveness in Schizophrenia Phase 1 Study. J Clin Psychiatry. 2020 Mar 17;81(2):19m12731. doi: 10.4088/JCP.19m12731. PMID 32220153
- [Derived] Ozzoude M, Nakajima S, Plitman E, Chung JK, Kim J, Iwata Y, Caravaggio F, Takeuchi H, Uchida H, Graff-Guerrero A, Gerretsen P. The effects of illness severity, cognition, and estimated antipsychotic dopamine receptor occupancy on insight into the illness in schizophrenia: An analysis of clinical antipsychotic trials of intervention effectiveness (CATIE) data. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:207-213. doi: 10.1016/j.pnpbp.2018.08.033. Epub 2018 Aug 30. PMID 30172739
- [Derived] Van Dyke P, Thomas KL. Concomitant calcium channel blocker and antipsychotic therapy in patients with schizophrenia: Efficacy analysis of the CATIE-Sz phase 1 data. Ann Clin Psychiatry. 2018 Feb;30(1):6-16. PMID 29069114
- [Derived] Xavier RM, Pan W, Dungan JR, Keefe RSE, Vorderstrasse A. Unraveling interrelationships among psychopathology symptoms, cognitive domains and insight dimensions in chronic schizophrenia. Schizophr Res. 2018 Mar;193:83-90. doi: 10.1016/j.schres.2017.07.002. Epub 2017 Jul 8. PMID 28693755
- [Derived] Bahorik AL, Greeno CG, Cochran G, Cornelius JR, Eack SM. Motivation deficits and use of alcohol and illicit drugs among individuals with schizophrenia. Psychiatry Res. 2017 Jul;253:391-397. doi: 10.1016/j.psychres.2017.04.012. Epub 2017 Apr 5. PMID 28441618
- [Derived] Moodie EE, Karran JC, Shortreed SM. A case study of SMART attributes: a qualitative assessment of generalizability, retention rate, and trial quality. Trials. 2016 May 14;17(1):242. doi: 10.1186/s13063-016-1368-3. PMID 27180047
- [Derived] Jakubovski E, Carlson JP, Bloch MH. Prognostic subgroups for remission, response, and treatment continuation in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) trial. J Clin Psychiatry. 2015 Nov;76(11):1535-45. doi: 10.4088/JCP.14m09320. PMID 26581028
- [Derived] Takeuchi H, Fervaha G, Remington G. Effect of Antipsychotic Dosing Regimen on Neurocognition in Schizophrenia. J Clin Psychopharmacol. 2015 Dec;35(6):728-30. doi: 10.1097/JCP.0000000000000424. No abstract available. PMID 26479222
- [Derived] Fervaha G, Agid O, Takeuchi H, Lee J, Foussias G, Remington G. Relationship between symptomatic improvement and overall illness severity in patients with schizophrenia. J Clin Psychopharmacol. 2015 Apr;35(2):128-33. doi: 10.1097/JCP.0000000000000286. PMID 25679125
- [Derived] Fervaha G, Agid O, Takeuchi H, Foussias G, Lee J, Remington G. Clinical and functional outcomes in people with schizophrenia with a high sense of well-being. J Nerv Ment Dis. 2015 Mar;203(3):187-93. doi: 10.1097/NMD.0000000000000266. PMID 25668654
- [Derived] Fervaha G, Takeuchi H, Lee J, Foussias G, Fletcher PJ, Agid O, Remington G. Antipsychotics and amotivation. Neuropsychopharmacology. 2015 May;40(6):1539-48. doi: 10.1038/npp.2015.3. Epub 2015 Jan 8. PMID 25567425
- [Derived] Fervaha G, Takeuchi H, Agid O, Lee J, Foussias G, Remington G. Determinants of patient-rated and clinician-rated illness severity in schizophrenia. J Clin Psychiatry. 2015 Jul;76(7):924-30. doi: 10.4088/JCP.14m09128. PMID 25562591
- [Derived] Fervaha G, Zakzanis KK, Foussias G, Graff-Guerrero A, Agid O, Remington G. Motivational deficits and cognitive test performance in schizophrenia. JAMA Psychiatry. 2014 Sep;71(9):1058-65. doi: 10.1001/jamapsychiatry.2014.1105. PMID 25075930
- [Derived] Marques TR, Levine SZ, Reichenberg A, Kahn R, Derks EM, Fleischhacker WW, Rabinowitz J, Kapur S. How antipsychotics impact the different dimensions of Schizophrenia: a test of competing hypotheses. Eur Neuropsychopharmacol. 2014 Aug;24(8):1279-88. doi: 10.1016/j.euroneuro.2014.04.001. Epub 2014 Apr 24. PMID 24862257
- [Derived] Fervaha G, Foussias G, Agid O, Remington G. Motivational and neurocognitive deficits are central to the prediction of longitudinal functional outcome in schizophrenia. Acta Psychiatr Scand. 2014 Oct;130(4):290-9. doi: 10.1111/acps.12289. Epub 2014 May 22. PMID 24850369
- [Derived] Fervaha G, Agid O, Takeuchi H, Foussias G, Remington G. Effect of antipsychotic medication on overall life satisfaction among individuals with chronic schizophrenia: findings from the NIMH CATIE study. Eur Neuropsychopharmacol. 2014 Jul;24(7):1078-85. doi: 10.1016/j.euroneuro.2014.03.001. Epub 2014 Mar 15. PMID 24726579
- [Derived] Fervaha G, Foussias G, Siddiqui I, Agid O, Remington G. Abbreviated quality of life scales for schizophrenia: comparison and utility of two brief community functioning measures. Schizophr Res. 2014 Apr;154(1-3):89-92. doi: 10.1016/j.schres.2014.02.013. Epub 2014 Mar 11. PMID 24630140
- [Derived] Witt K, Hawton K, Fazel S. The relationship between suicide and violence in schizophrenia: analysis of the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) dataset. Schizophr Res. 2014 Apr;154(1-3):61-7. doi: 10.1016/j.schres.2014.02.001. Epub 2014 Feb 26. PMID 24581550
- [Derived] Takeuchi H, Fervaha G, Uchida H, Suzuki T, Bies RR, Gronte D, Remington G. Impact of once- versus twice-daily perphenazine dosing on clinical outcomes: an analysis of the CATIE data. J Clin Psychiatry. 2014 May;75(5):506-11. doi: 10.4088/JCP.13m08695. PMID 24569099
- [Derived] Bahorik AL, Newhill CE, Queen CC, Eack SM. Letter to the editor: Critique of Bahorik et al. (2013)--'Underreporting of drug use among individuals with schizophrenia: prevalence and predictors'--a reply. Psychol Med. 2014 Feb;44(3):670-1. doi: 10.1017/s0033291713002560. No abstract available. PMID 24524169
- [Derived] Laber EB, Lizotte DJ, Ferguson B. Set-valued dynamic treatment regimes for competing outcomes. Biometrics. 2014 Mar;70(1):53-61. doi: 10.1111/biom.12132. Epub 2014 Jan 8. PMID 24400912
- [Derived] Fervaha G, Agid O, Takeuchi H, Foussias G, Remington G. Clinical determinants of life satisfaction in chronic schizophrenia: data from the CATIE study. Schizophr Res. 2013 Dec;151(1-3):203-8. doi: 10.1016/j.schres.2013.10.021. Epub 2013 Nov 1. PMID 24183751
- [Derived] Fervaha G, Agid O, Takeuchi H, Foussias G, Remington G. Life satisfaction among individuals with schizophrenia in the Clinical Antipsychotic Trial of Intervention Effectiveness (CATIE) study. Am J Psychiatry. 2013 Sep;170(9):1061-2. doi: 10.1176/appi.ajp.2013.13010060. No abstract available. PMID 24030617
- [Derived] Takeuchi H, Suzuki T, Bies RR, Remington G, Mamo DC, Pollock BG, Mimura M, Uchida H. Estimated dopamine D2 receptor occupancy from plasma concentrations of atypical antipsychotics and subjective experience/drug attitude in schizophrenia: an analysis of the CATIE data. Schizophr Res. 2013 Nov;150(2-3):373-9. doi: 10.1016/j.schres.2013.08.033. Epub 2013 Sep 9. PMID 24028745
- [Derived] Tsuboi T, Bies RR, Suzuki T, Mamo DC, Pollock BG, Graff-Guerrero A, Mimura M, Uchida H. Hyperprolactinemia and estimated dopamine D2 receptor occupancy in patients with schizophrenia: analysis of the CATIE data. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Aug 1;45:178-82. doi: 10.1016/j.pnpbp.2013.05.010. Epub 2013 May 29. PMID 23727135
- [Derived] Fervaha G, Remington G. Validation of an abbreviated quality of life scale for schizophrenia. Eur Neuropsychopharmacol. 2013 Sep;23(9):1072-7. doi: 10.1016/j.euroneuro.2012.11.009. Epub 2012 Dec 9. PMID 23235268
- [Derived] Levine SZ, Rabinowitz J, Faries D, Lawson AH, Ascher-Svanum H. Treatment response trajectories and antipsychotic medications: examination of up to 18 months of treatment in the CATIE chronic schizophrenia trial. Schizophr Res. 2012 May;137(1-3):141-6. doi: 10.1016/j.schres.2012.01.014. Epub 2012 Feb 7. PMID 22316567
- [Derived] Sakurai H, Bies RR, Stroup ST, Keefe RS, Rajji TK, Suzuki T, Mamo DC, Pollock BG, Watanabe K, Mimura M, Uchida H. Dopamine D2 receptor occupancy and cognition in schizophrenia: analysis of the CATIE data. Schizophr Bull. 2013 May;39(3):564-74. doi: 10.1093/schbul/sbr189. Epub 2012 Jan 30. PMID 22290266
- [Derived] Levine SZ, Rabinowitz J, Ascher-Svanum H, Faries DE, Lawson AH. Extent of attaining and maintaining symptom remission by antipsychotic medication in the treatment of chronic schizophrenia: evidence from the CATIE study. Schizophr Res. 2011 Dec;133(1-3):42-6. doi: 10.1016/j.schres.2011.09.018. Epub 2011 Oct 14. PMID 22000938
- [Derived] Addington DE, Mohamed S, Rosenheck RA, Davis SM, Stroup TS, McEvoy JP, Swartz MS, Lieberman JA. Impact of second-generation antipsychotics and perphenazine on depressive symptoms in a randomized trial of treatment for chronic schizophrenia. J Clin Psychiatry. 2011 Jan;72(1):75-80. doi: 10.4088/JCP.09m05258gre. Epub 2010 Sep 21. PMID 20868641
- [Derived] Caroff SN, Davis VG, Miller DD, Davis SM, Rosenheck RA, McEvoy JP, Campbell EC, Saltz BL, Riggio S, Chakos MH, Swartz MS, Keefe RS, Stroup TS, Lieberman JA; CATIE Investigators. Treatment outcomes of patients with tardive dyskinesia and chronic schizophrenia. J Clin Psychiatry. 2011 Mar;72(3):295-303. doi: 10.4088/JCP.09m05793yel. Epub 2010 Aug 10. PMID 20816031
- [Derived] Meyer JM, McEvoy JP, Davis VG, Goff DC, Nasrallah HA, Davis SM, Hsiao JK, Swartz MS, Stroup TS, Lieberman JA. Inflammatory markers in schizophrenia: comparing antipsychotic effects in phase 1 of the clinical antipsychotic trials of intervention effectiveness study. Biol Psychiatry. 2009 Dec 1;66(11):1013-22. doi: 10.1016/j.biopsych.2009.06.005. Epub 2009 Jul 29. PMID 19640511